CLINICAL TRIAL: NCT03530111
Title: Establishment of the 2H-labeling Protocol to Assess in Vivo Adipose Tissue Dynamics at PBRC
Brief Title: Establishment of the 2H-labeling Protocol at Pennington Biomedical Research Center
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Ursula White, Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2018-004
Record Dates: First submitted 2018-05-02; First posted 2018-05-21 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Overweight and Obesity; Exercise
Keywords: Adipose tissue; Adipose turnover; Adipose kinetics; Exercise; Deuterium
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Adipose tissue biopsies from the subcutaneous abdominal and femoral regions will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sedentary: Sedentary individuals will be classified as achieving < 75 minutes of moderate-intensity or < 37 minutes of vigorous-intensity aerobic physical activity per week.
- Very Physically Active: Very Physically Active individuals will be classified as achieving > 225 minutes of moderate-intensity or > 112 minutes of vigorous-intensity aerobic physical activity per week.

SUMMARY:
A method has been developed to measure in vivo adipose kinetics and turnover rates, which is a substantive departure from previous indirect and in vitro approaches. This technique involves drinking deuterium (2H)-labeled water, with an initial ramp-up to increase body water 2H enrichment, followed by daily intake to maintain enrichment values. The 2H from the heavy water is incorporated into the DNA of the dividing cells, as well as the lipid component, providing measures of cell formation, lipid synthesis, and adipose turnover. The objective of the proposed study is to enroll women who are overweight (sedentary or physically active) in order to collect 2H-enriched adipose tissue specimens that will be utilized to establish this innovative 2H-labeling protocol at Pennington Biomedical Research Center. This study will also assess adipose kinetics in individuals with different levels of physical activity to better understand the association between in vivo adipose cell kinetics, physical activity, and metabolic health in humans.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women
* 18-40 years of age
* BMI 25-29.9 kg/m2 (+/- 0.5 will be accepted)
* Are willing to drink deuterium-labeled water (2H2O) for 6 weeks
* Must be willing to comply with all study procedures, including adipose biopsies and a DXA scan
* If applicable, hormonal contraception must have been started at least 2 months before entering the study. If enrolled, subject must also agree to not alter hormonal birth control method, dose, or regimen throughout the duration of the study
* If not using pharmaceutical (hormonal) contraception (i.e. birth control pills, vaginal ring, injections, or implant), agree to use a double barrier method as a form of birth control to prevent pregnancy
* Must be classified as either sedentary (achieve < 75 minutes of moderate-intensity or < 37 minutes of vigorous-intensity aerobic physical activity per week) or very physically active (achieve > 225 minutes of moderate-intensity or > 112 minutes of vigorous-intensity aerobic physical activity per week). Simple questions to assess physical activity level will be administered during the phone screening as well as the clinic screening visit.
* If enrolled, agree to not alter dose, level, or regimen of physical activity throughout the duration of the study

Exclusion Criteria:

* Unstable weight in the last 3 months (gain or loss >7 lb (3.2 kg)
* Significant changes in the diet or level of physical activity within the past month
* History of clinically diagnosed diabetes or a fasting blood glucose > 110 mg/dL
* An average screening blood pressure >140/90
* Have major organ disease (i.e. heart, kidney, lung, thyroid, or liver) or abnormal liver enzymes that are, in the opinion of the medical investigator, clinically significant and represent a problem for study inclusion.
* Self-reported positive test for human immunodeficiency virus, hepatitis B and hepatitis C
* Chronic use of systemic glucocorticoids, systemic adrenergic-stimulating agents, anti-psychotic/anti-depressant medications, thiazolidinediones and other medications that may cause clinically significant weight gain or loss
* Chronic use of prescription or over-the-counter weight loss medications which, in the opinion of the MI, will impact the study.
* Smoking or use of tobacco products in the last 3 months
* Pregnancy, breastfeeding, or planned pregnancy for the upcoming 2 months
* Previous bariatric or other surgeries for obesity
* Diagnosed psychotic conditions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 12 women who are overweight and are either sedentary or very physically active will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Measures (fractional synthesis) of In vivo Adipose Cell Formation | 1 year
  Following the consumption of deuterium-labeled water (2H2O; heavy water), adipose tissue biopsies from the subcutaneous abdominal and femoral depots will be collected. The 2H from the heavy water is enriched into the DNA of newly synthesized cells. Measures of DNA synthesis (obtained via gas chromatography and mass spectrometry analysis of 2H-enrichment) denote new adipose cell formation. The primary outcome is to assess adipose cell kinetic rates (i.e. synthesis) in sedentary and very physically active women.

SECONDARY OUTCOMES:
Measures (fractional synthesis) of In vivo Triglyceride Synthesis | 1 year
  Following the consumption of deuterium-labeled water (2H2O; heavy water), adipose tissue biopsies from the subcutaneous abdominal and femoral depots will be collected. The 2H from the heavy water is incorporated into the glycerol component of the adipose, providing a measure of new triglyceride synthesis. The secondary outcome is to assess adipose lipid (triglyceride) kinetic rates (i.e. synthesis) in sedentary and very physically active women.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula White, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided